CLINICAL TRIAL: NCT07295756
Title: The Role of Smoking Habits in Periodontal Health and Disease: A Cross-Sectional Study
Brief Title: The Role of Smoking in Periodontal Status
Acronym: TRSPS
Status: Completed | Type: Observational
Sponsor: Tuğba ŞAHİN (Other)
Responsible Party: Sponsor-Investigator, Tuğba ŞAHİN, Assistant professor, Abant Izzet Baysal University
Organization: Abant Izzet Baysal University (Other)
Other Study IDs: BAIBU-DH-TS-05
Record Dates: First submitted 2025-11-18; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Periodontal Diseases
Keywords: periodontal diseases; periodontitis; smoking; gingivitis; tabocco products
MeSH Terms: conditions — Periodontal Diseases; Periodontitis; Smoking; Gingivitis | interventions — Methods; Smoking Devices

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Smoker: Current smokers were defined as individuals who had smoked ≥100 cigarettes in their lifetime and continued smoking.
  Interventions: Other: Intervention
- Non-smoker: Non-smokers included individuals who had smoked fewer than 100 cigarettes in their lifetime and were not currently smoking.
  Interventions: Other: Intervention

INTERVENTIONS:
Other: Intervention — The patient's daily cigarette consumption, duration of smoking, and pack-years were evaluated.
  Other Names: Smoking

SUMMARY:
484 patients were asked whether they currently smoked and whether they had smoked 100 or more cigarettes during their lifetime. Based on this information, they were divided into two groups: current smokers (test group, n=242) and non-smokers (control group, n=242). Current smokers were defined as individuals who had smoked ≥100 cigarettes in their lifetime and continued smoking. In contrast, non-smokers included individuals who had smoked fewer than 100 cigarettes in their lifetime and were not currently smoking. Participants were also asked about the number of cigarettes smoked per day and the duration of smoking in years, and pack-years were calculated accordingly. Plaque index, gingival index, probing depth, bleeding on probing, gingival recession, and attachment loss were evaluated for both groups. Periodontal health status (Periodontal health, gingivitis, and periodontitis) was assessed by one clinician applying the 2017 World Workshop on Classifying Periodontal and Peri-Implant Diseases and Conditions and the 2023 European Federation of Periodontology's Guidelines. Patients with periodontitis were classified according to stage and grade. This measurement was obtained via a calibrated UNC-15 periodontal probe at each tooth.

DETAILED DESCRIPTION:
484 patients were asked whether they currently smoked and had smoked 100 or more cigarettes during their lifetime. Based on this information, they were divided into two groups: current smokers (test group, n=242) and non-smokers (control group, n=242). Current smokers were defined as individuals who had smoked ≥100 cigarettes in their lifetime and continued smoking. In contrast, non-smokers included individuals who had smoked fewer than 100 cigarettes in their lifetime and were not currently smoking. Participants were also asked about the number of cigarettes smoked per day and the duration of smoking in years, and pack-years were calculated accordingly. Plaque index, gingival index, probing depth, bleeding on probing, gingival recession, and attachment loss were evaluated for both groups. Periodontal health status (Periodontal health, gingivitis, and periodontitis) was assessed by one clinician applying the 2017 World Workshop on Classifying Periodontal and Peri-Implant Diseases and Conditions and the 2023 European Federation of Periodontology's Guidelines. Patients with periodontitis were classified according to stage and grade. This measurement was obtained via a calibrated UNC-15 periodontal probe at each tooth.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* No systemic diseases that could affect periodontal or general health
* No history of periodontal treatment within the past six months
* For the non-smoker group: abstinence from smoking for at least five years

Exclusion Criteria:

* Use of antibiotics or anti-inflammatory drugs
* Pregnant or lactating women
* Diabetes mellitus
* Use of waterpipe or chewing tobacco (for the smoker group)
* Individuals undergoing chemotherapy or radiotherapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study includes patients who are smokers and those who are non-smokers.
Sampling Method: Non-Probability Sample
Enrollment: 484 (Actual)
Dates: Start 2025-01-02 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2025-10-02 (Actual)

PRIMARY OUTCOMES:
periodontal pocket depth | Baseline
  Periodontal pocket depth measured in millimeters using a Williams periodontal probe. The distance from the gingival margin to the bottom of the periodontal pocket was recorded at each site.

SECONDARY OUTCOMES:
bleeding on probing | Baseline
  Bleeding on probing assessed using a periodontal probe. After gently inserting the probe into the gingival sulcus and moving it laterally along the pocket wall, bleeding was recorded as present (+) or absent (-).pocket and gently moved laterally along the pocket wall. + is maximum and - is minimum.
plaque index | Baseline
  Oral hygiene status assessed using the Plaque Index, which measures dental plaque accumulation adjacent to the gingival margin. Scores range from 0 (no plaque) to 3 (abundant plaque), with higher scores indicating poorer oral hygiene.
gingival index | Baseline
  Gingival inflammation assessed using the Löe and Silness Gingival Index. Each site was scored on a 0-3 scale, where 0 = normal gingiva and 3 = severe inflammation with edema, redness, and spontaneous bleeding. Higher scores indicate worsening gingival inflammation.
clinical attachment level | Baseline
  Clinical attachment level measured in millimeters using a periodontal probe. CAL was calculated as the distance from the cementoenamel junction to the bottom of the periodontal pocket and used to assess periodontal tissue support loss.
Daily cigarette | Baseline
  It includes the number of cigarettes smoked per day. Self-reported number of cigarettes smoked per day.
Smoking Duration | Baseline
  Self-reported duration of smoking, recorded as the number of years the participant has smoked.
Pack-years | Baseline
  Smoking exposure calculated as pack-years, defined as the number of cigarettes smoked per day divided by 20 and multiplied by the number of years of smoking.

CONTACTS AND LOCATIONS:
Overall Officials: TUGBA SAHIN, Principal Investigator — Abant Izzet Baysal University
Locations (1):
- Bolu Abant Izzet Baysal University, Dentistry Faculty, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided